CLINICAL TRIAL: NCT01573767
Title: A Dose-ranging Study of Vilanterol (VI) Inhalation Powder in Children Aged 5-11 Years With Asthma on a Background of Inhaled Corticosteroid Therapy
Brief Title: Dose-ranging Study of Vilanterol (VI) Inhalation Powder in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 106853
Record Dates: First submitted 2012-03-08; First posted 2012-04-10 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): Vilanterol 25mcg inhalation powder inhaled once daily in the PM via the new powder inhaler
  Interventions: Drug: Fluticasone propionate 100mcg; Drug: Vilanterol
- Arm 2 (Active Comparator): Vilanterol 12.5mcg inhalation powder inhaled once daily in the PM via the new powder inhaler
  Interventions: Drug: Fluticasone propionate 100mcg; Drug: Vilanterol
- Arm 3 (Active Comparator): Vilanterol 6.25mcg inhalation powder inhaled once daily in the PM via the new powder inhaler
  Interventions: Drug: Fluticasone propionate 100mcg; Drug: Vilanterol
- Arm 4 (Placebo Comparator): Placebo inhalation powder inhaled once daily in the PM via the new powder inhaler
  Interventions: Drug: Fluticasone propionate 100mcg; Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate 100mcg — all subjects recieve open-label Flovent twice daily duirng the run in and treatment period
Drug: Placebo — Placebo inhalation powder during treatment period
  Arms: Arm 4
Drug: Vilanterol — subjects will recieve 4 weeks via NDPI during treament period
  Arms: Arm 1; Arm 2; Arm 3

SUMMARY:
This is a Phase IIb, multi-centre, randomised, double-blind, parallel-group, placebo-controlled study in children aged 5-11 years with persistent uncontrolled asthma. Subjects entering the run-in period will stop their current asthma medication and be given open label fluticasone propionate (FP) 100mcg twice daily via DISKUS/ACCUHALER and salbutamol/albuterol as required to use throughout the run-in and double-blind treatment period. At Visit 3 subjects meeting the randomization eligibility criteria will receive vilanterol (6.25mcg, 12.5mcg, or 25mcg,) or placebo via the Novel Dry Powder Inhaler (NDPI) once daily for 4 weeks in addition to open-label fluticasone propionate twice daily throughout the treatment period. Primary endpoints consist of change from baseline in clinic visit trough (pre-bronchodilator and pre-dose) PEF at the end of the 28-day treatment period in all subjects. Safety assessments include adverse events, oropharyngeal examinations, clinical chemistry, 12-lead ECG, and vital signs. Blood samples will be taken from all subjects for pharmacokinetic analysis to determine plasma concentrations of vilanterol at specific time intervals relative to the dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from at least one parent/ legal guardian to take part in the study.:
* Diagnosis of asthma
* pre-bronchodilator PEF between ≥50% to ≤90% of their best post-bronchodilator value
* Receiving stable asthma therapy of short acting beta-agonist (SABA) plus ICS (total daily dose FP 200mcg or equivalent)

Exclusion Criteria:

* history of life-threatening asthma
* history of asthma exacerbation for asthma within 6 months prior to screening.
* Culture-documented or suspected bacterial or viral infection
* significant abnormality or medical condition
* Present use of any tobacco products

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 463 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (106):
- United States (34):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Shiloh, Illinois
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Nicholasville, Kentucky
  - GSK Investigational Site, White Marsh, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Spring, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
- Argentina (12):
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, San Juan Bautista, Buenos Aires
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Salta, Salta Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (4):
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Viña del Mar
- GSK Investigational Site, Tbilisi, Georgia
- Germany (17):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Baunatal-Grossenritte, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Hamm, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Wesel, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Neuhaus am Rennweg, Thuringia
- Japan (8):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
- Mexico (4):
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Puebla, Pue, Puebla
  - GSK Investigational Site, Villahermosa, Tabasco
  - GSK Investigational Site, Mexico City
- Peru (3):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Santiago de Surco, Lima region
- Philippines (3):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (9):
  - GSK Investigational Site, Bieńkówka
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Oleśnica
  - GSK Investigational Site, Ostrów Wielkopolski
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zawadzkie
- GSK Investigational Site, Hato Rey, Puerto Rico, Puerto Rico
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Vysoké Tatry
- South Africa (4):
  - GSK Investigational Site, Meyerspark, Gauteng
  - GSK Investigational Site, CapeTown
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Panorama
- Ukraine (3):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Oliver AJ, Covar RA, Goldfrad CH, Klein RM, Pedersen SE, Sorkness CA, Tomkins SA, Villaran C, Grigg J. Randomised trial of once-daily vilanterol in children with asthma on inhaled corticosteroid therapy. Respir Res. 2016 Apr 5;17:37. doi: 10.1186/s12931-016-0353-4. PMID 27044326
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1208 participants (par.) were screened; 760 entered the Run-in Phase, 463 were randomized, and 2 received study medication (SM) but weren't randomized/included in the Intent-to-Treat (ITT) Population (randomized to treatment and receiving >=1 SM dose). 7 randomized par. didn't receive SM; hence, 456 par. comprised the ITT Population.
Pre-assignment Details: Participants who met the eligibility criteria at screening (Visit 1) entered the Run-in Phase for completion of Baseline safety evaluations and measures of asthma status. Participants meeting all randomization criteria at Visit 3 were randomized to 1 of 4 treatment arms. The total duration of study participation was up to a maximum of 9 weeks.
Groups:
- Placebo: Participants received placebo once daily (OD) in the evening from a dry powder inhaler for 4 weeks in addition to open-label fluticasone propionate (FP) 100 micrograms (µg) twice daily (BID). Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
- VI 6.25 µg OD: Participants received vilanterol (VI) 6.25 µg OD in the evening from a dry powder inhaler for 4 weeks in addition to open-label FP 100 µg BID. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
- VI 12.5 µg OD: Participants received VI 12.5 µg OD in the evening from a dry powder inhaler for 4 weeks in addition to open-label FP 100 µg BID. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
- VI 25 µg OD: Participants received VI 25 µg OD in the evening from a dry powder inhaler for 4 weeks in addition to open-label FP 100 µg BID. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
Period: Overall Study
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Started | 115 | 114 | 113 | 114
Completed | 93 | 93 | 99 | 90
Not Completed | 22 | 21 | 14 | 24
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Lack of Efficacy | 18 | 15 | 12 | 17
Not completed — Protocol Violation | 3 | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD | Total
Number analyzed (Participants) | 115 | 114 | 113 | 114 | 456
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (1.81) | 8.0 (1.95) | 7.9 (1.74) | 7.9 (1.72) | 7.9 (1.80)
Gender [Count of Participants; unit: Participants]
  Female | 50 | 43 | 42 | 45 | 180
  Male | 65 | 71 | 71 | 69 | 276
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 5 | 5 | 5 | 3 | 18
  American Indian or Alaska Native | 16 | 21 | 17 | 18 | 72
  Asian - Japanese Heritage | 5 | 5 | 5 | 5 | 20
  Asian - South East Asian Heritage | 1 | 1 | 2 | 1 | 5
  White - Arabic/North African Heritage | 1 | 1 | 0 | 1 | 3
  White - White/Caucasian/European Heritage | 67 | 62 | 55 | 61 | 245
  Mixed Race | 20 | 19 | 29 | 25 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Pre-dose Evening (PM) Peak Expiratory Flow (PEF) From Participant Electronic Daily Diary Averaged Over the 4-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use each morning. The best of three measurements was recorded. Change from Baseline was calculated as the value of the averaged daily PM PEF over the 4-week Treatment Period minus the Baseline value. The Baseline PEF value is defined as the average of the last 7 days of the Run-in Phase. The analysis was performed using an analysis of covariance (ANCOVA) model with covariates of Baseline, region, sex, age, and treatment. Only those participants contributing data per the daily eDiary were analyzed.
Time Frame: Baseline; Week 1 up to Week 4
Population: ITT Population: participants randomized to treatment who received >=1 dose of study medication
Measure: Least Squares Mean (Standard Error); unit: Liters per minute (L/min)
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 113 | 113 | 112 | 110
Liters per minute (L/min) | 215.9 (2.53) | 221.4 (2.53) | 222.4 (2.54) | 220.3 (2.56)
Statistical Analysis 1: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; p = 0.227, ANCOVA — Inference for VI 12.5 µg versus (vs) placebo was dependent upon statistical significance (SS) having first been achieved for VI 25 µg vs placebo; inference for VI 6.25 µg vs placebo was dependent on SS having been achieved for VI 12.5 µg vs placebo; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [-2.7 to 11.4]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; p = 0.073, ANCOVA; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-0.6 to 13.5]
Statistical Analysis 3: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; p = 0.127, ANCOVA; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-1.6 to 12.5]

2. Secondary Outcome: Change From Baseline in Evening Clinic Visit Trough (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 4-week Treatment Period in Children Who Could Perform the Maneuver
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as a pre-dose FEV1 measurement taken at a clinic visit while still on treatment. Change from Baseline in trough FEV1 at the end of the 4-week Treatment Period was defined using the pre-dose FEV1 measurement taken at the Week 4 clinic visit. Change from Baseline was calculated as the Week 4 trough FEV1 value minus the Baseline value. The Baseline FEV1 value is defined as the value at Visit 3 (randomization). The analysis was performed using an ANCOVA model with covariates of Baseline trough FEV1, region, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing measurements.
Time Frame: Baseline; Week 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 85 | 83 | 86 | 86
Liters | 0.223 (0.0287) | 0.166 (0.0292) | 0.240 (0.0285) | 0.193 (0.0288)
Statistical Analysis 1: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.057, 95% CI 2-sided [-0.138 to 0.024]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.063 to 0.096]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.110 to 0.051]

3. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour Periods During the 4-week Treatment Period
Description: The number of inhalations of rescue albuterol/salbutamol inhalation aerosol (medication used to relieve symptoms immediately) used during the day and night) was recorded by the participants in a daily diary. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered as rescue free. Participants who were rescue free for 24-hour periods during the 4-week Treatment Period were assessed. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant. Change from Baseline is calculated as the average value during the 4-week Treatment Period minus the value at Baseline. The Baseline value is defined as the value at Visit 3 (randomization). Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline; Week 1 up to Week 4
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 113 | 113 | 112 | 110
Percentage of rescue-free 24-hr periods | 14.4 (2.97) | 12.2 (2.97) | 15.8 (2.98) | 2.98 (3.01)
Statistical Analysis 1: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-10.5 to 6.0]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-6.9 to 9.6]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [0.4 to 17.0]

4. Secondary Outcome: Change From Baseline in Daily Morning (AM) PEF Averaged Over the 4-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline was calculated as the value of the averaged daily AM PEF over the 4-week Treatment Period (at Week 4) minus the Baseline value. The Baseline value is defined as the value at Visit 3 (randomization). The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: Baseline; Week 1 up to Week 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 114 | 113 | 112 | 110
L/min | 6.4 (2.42) | 12.0 (2.43) | 13.9 (2.44) | 13.7 (2.46)
Statistical Analysis 1: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-1.2 to 12.3]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [0.7 to 14.2]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 7.2, 95% CI [0.4 to 14.0]

5. Secondary Outcome: Change From Baseline in Evening (PM) PEF Over the Last 7 Days of the Treatment Period (Week 4)
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline is calculated as the value over the last 7 days of the Treatment Period minus the Baseline value. The Baseline value is defined as the value at Visit 3 (randomization). The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing measurements.
Time Frame: Baseline; Week 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 113 | 113 | 112 | 110
L/min | 5.9 (3.44) | 9.4 (3.44) | 13.7 (3.45) | 11.1 (3.48)
Statistical Analysis 1: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-6.1 to 13.1]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-1.8 to 17.4]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-4.4 to 14.9]

6. Secondary Outcome: Change From Baseline in AM PEF Over the Last 7 Days of the Treatment Period (Week 4)
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline is calculated as the value of the averaged daily AM PEF over the 4-week Treatment Period (at Week 4) minus the Baseline value. The Baseline value is defined as the value at Visit 3 (randomization). The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: Baseline; Week 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 114 | 113 | 112 | 110
L/min | 7.4 (3.45) | 13.3 (3.47) | 17.0 (3.48) | 14.4 (3.51)
Statistical Analysis 1: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-3.7 to 15.6]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 9.7, 95% CI 2-sided [0.0 to 19.3]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 7.0, 95% CI [-2.7 to 16.7]

7. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour Periods During the 4-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the PEF measurement. A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. The Baseline symptom-free value is defined as the value at Visit 3 (randomization). Change from Baseline was calculated as the averaged value during the 4-week Treatment Period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment group.
Time Frame: Baseline; Week 1 up to Week 4
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | VI 6.25 µg OD | VI 12.5 µg OD | VI 25 µg OD
Number analyzed (Participants) | 113 | 113 | 112 | 110
Percentage of symptom-free 24-hr periods | 9.9 (2.65) | 10.1 (2.65) | 18.3 (2.66) | 19.7 (2.69)
Statistical Analysis 1: Comparison: Placebo vs VI 6.25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-7.2 to 7.5]
Statistical Analysis 2: Comparison: Placebo vs VI 12.5 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [1.0 to 15.7]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [2.3 to 17.2]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the follow-up visit (up to 9 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants who were randomized to treatment and received at least one dose of study medication.
Groups:
- VI 6.25 OD: Participants received vilanterol (VI) 6.25 µg OD in the evening from a dry powder inhaler for 4 weeks in addition to open-label FP 100 µg BID. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
- VI 12.5 OD: Participants received VI 12.5 µg OD in the evening from a dry powder inhaler for 4 weeks in addition to open-label FP 100 µg BID. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
- VI 25 OD: Participants received VI 25 µg OD in the evening from a dry powder inhaler for 4 weeks in addition to open-label FP 100 µg BID. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication.
Arm/Group | Placebo | VI 6.25 OD | VI 12.5 OD | VI 25 OD
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/114 | 0/113 | 1/114
Other Adverse Events (participants affected / at risk) | 10/115 | 17/114 | 12/113 | 11/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | VI 6.25 OD (N=114) | VI 12.5 OD (N=113) | VI 25 OD (N=114)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | VI 6.25 OD (N=114) | VI 12.5 OD (N=113) | VI 25 OD (N=114)
Nasopharyngitis (Infections and infestations) | 8 | 8 | 10 | 9
Influenza (Infections and infestations) | 0 | 4 | 0 | 0
Headache (Nervous system disorders) | 4 | 6 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.